CLINICAL TRIAL: NCT06727994
Title: The Effect of Genital Hygiene Education on the Self-Care Agency and Genital Hygiene Behaviors of Incarcerated Women
Brief Title: Genital Hygiene Education of Incarcerated Women
Acronym: GHEIW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Hüsne YÜCESOY, PhD, Ordu University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Ordu Üniversitesi
Record Dates: First submitted 2024-05-24; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Genital Hygiene

STUDY DESIGN:
Intervention Model Description: The studyis of a semi-separate typeand all women can be trained
Masking Description: The studyis of a semi-separate typeand all women can be trained
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- training group (Experimental): Providing Genital Hygiene training
  Interventions: Other: Providing Genital Hygiene training

INTERVENTIONS:
Other: Providing Genital Hygiene training — After the informed consent of all participants in the study is obtained, pre-test data, Self-Care Power Scale and Genital Hygiene Behavior Scale will be collected face-to-face.
  "Genital Hygiene" training will be given. Reminder training will be given 15 days, 1 month and 2 months after the training, and 1 month after the reminder training, the Self-Care Power Scale and Genital Hygiene Behavior Scale will be re-administered to women as a final test.

SUMMARY:
Pretest data will be collected after obtaining informed consent from all study participants. Pre-test data will be collected using the Personal Information Form, Self-Care Strength Scale and Genital Hygiene Behavior Scale. Genital Hygiene training will be given after pre-test data is collected. Reminder training will be given after the first training. Reminder training will be given 15 days, 1 month and 2 months after the training. Post-test data will be collected 1 month after the last reminder training. Post-test data will be collected using the Self-Care Strength Scale and Genital Hygiene Behavior Scale.

DETAILED DESCRIPTION:
Type of research The research was planned as a quasi-experimental and was planned in a pre-test post-test grouped order.

Population and sample of the research The population of the research consists of 70 female prisoners in Çorum L-type Closed Penal Institution. Considering the benefit of the study to all women, all female prisoners who agree to participate in the research and meet the inclusion criteria, without any sample selection, will constitute the sample of the quasi-experimental study.

Collection of research data The data of the research will be collected from the prisoners in the women's unit of the relevant Penal Institution. Personal Information Form, Self-Care Power Scale and Genital Hygiene Behavior Scale will be used to collect research data.

Personal Information Form: It consists of questions regarding women's sociodemographic characteristics and genital discharge status.

Self-Care Power Scale: The scale is a tool developed by Kearney and Fleischer in 1979 to determine individuals' ability and strength to take care of themselves (Kearney and Fleischer, 1979). The validity and reliability study of the scale was conducted by Nakhcivan in Turkey in 1993 (Nahcivan, 1994). The scale consists of 35 items that aim to evaluate individuals' self-care abilities and strengths and is a 5-point Likert type. The maximum score to be obtained from the scale is 140, below 82 points is considered low, 82-120 points is considered medium, and above 120 points is considered high self-care ability. An increase in the score obtained from the scale indicates that the individual's self-care power increases. The Cronbach's alpha value of the original scale is 0.89.

Genital Hygiene Behaviors Scale (GHDS): The Genital Hygiene Behaviors Scale, which was developed and validated by Karahan in 2017, is in Likert type. It is rated from 5 to 1, from "I completely agree" to "I completely disagree", and it consists of 23 statements. The scale has three sub-dimensions: general hygiene (first 12 items), menstrual hygiene (items 13-20) and awareness of abnormal findings (items 21-23). In evaluating the scale, items 7, 14, 19, 20, 23 are reverse coded; The lowest score from the scale can be 23 and the highest score can be 115, and it shows that women with high scores have good genital hygiene behavior (Karahan, 2017). The Cronbach's alpha value of the original scale is 0.80.

Protocol of the Research After the informed consent of all participants in the study is obtained, pre-test data will be collected face-to-face with the Personal Information Form, Self-Care Power Scale and Genital Hygiene Behavior Scale.

The training will include information about vaginal discharge and its characteristics, common genital infections, wrong behaviors and practices that cause vaginal infections, the importance of genital infections for women's health, and correct genital hygiene behaviors.

"Genital Hygiene" training will be given. Reminder training will be given 15 days, 1 month and 2 months after the training, and 1 month after the reminder training, the Self-Care Power Scale and Genital Hygiene Behavior Scale will be re-administered to women as a final test.

Estimated completion time of the research: 6 months. Criteria for inclusion in the study

* Volunteering to participate in the study,
* Being between the ages of 18-65,
* To know Turkish. Exclusion criteria from the study
* Not attending employee training regularly,
* Leaving the study in the later stages of the study.

Statistical analysis methods to be used Data analysis of the study will be carried out in a computer environment using the SPSS 21.0 program. Descriptive statistics including number, percentage, standard deviation and parametric or non-parametric analysis tests will be used depending on the normal distribution of the data. For repeated tests, paired sample test will be applied in parametric groups. A value of p≤0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study,
* Being between the ages of 18-65,
* To know Turkish.

Exclusion Criteria:

* Not attending employee training regularly,
* Leaving the study in the later stages of the study.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — suitable
Enrollment: 70 (Actual)
Dates: Start 2024-05-20 (Actual); Primary Completion 2024-07-20 (Actual); Study Completion 2024-09-20 (Actual)

PRIMARY OUTCOMES:
The Effect of Genital Hygiene Education on the Self-Care Agency and Genital Hygiene Behaviors of Incarcerated Women | one months
  preliminary test results
  Genital Hygiene Behaviors Scale (GHDÖ): The Genital Hygiene Behaviors Scale, which was developed by Karahan in 2017 and whose validity and reliability were conducted, is a Likert-type scale. It is graded from 5 to 1 from "I completely agree" to "I completely disagree" and consists of 23 statements. The scale has three sub-dimensions: general hygiene (first 12 items), menstrual hygiene (items 13-20), and abnormal finding awareness (items 21-23). In the evaluation of the scale, items 7, 14, 19, 20, and 23 are reverse-coded; the lowest score can be obtained from the scale is 23 and the highest is 115, and women with high scores show that their genital hygiene behavior is good (Karahan, 2017). The Cronbach alpha value of the original scale is 0.80.

SECONDARY OUTCOMES:
The Effect of Genital Hygiene Education on the Self-Care Agency and Genital Hygiene Behaviors of Incarcerated Women | 3 months
  final test results
  Self-Care Abilities Scale: The scale is a tool developed by Kearney and Fleischer in 1979 to determine the ability and strength of individuals to care for themselves (Kearney and Fleischer, 1979). The validity and reliability study of the scale was conducted by Nahcivan in Turkey in 1993 (Nahcivan, 1994). The scale consists of 35 items that aim to evaluate the ability and strength of individuals to care for themselves and is a 5-point Likert-type scale. The maximum score that can be obtained from the scale is 140, and below 82 points is considered low, 82-120 points is considered medium, and above 120 points is considered high self-care ability. An increase in the score obtained from the scale indicates that the individual's self-care ability increases. The Cronbach alpha value of the original scale is 0.89.

CONTACTS AND LOCATIONS:
Overall Officials: husne yucesoy, Principal Investigator — ordu üniversitesi
Locations (2):
- Turkey (Türkiye) (2):
  - Ordu Üniversitesi, Ordu, Altınordu
  - Ordu Üniversitesi, Ordu